CLINICAL TRIAL: NCT05292196
Title: A Randomized, Double-blind, Placebo-parallel, Multicenter Phase II Trial of the Efficacy and Safety of TQC3721 Suspension for Inhalation in the Treatment of Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Phase II Clinical Trial of TQC3721 Suspension for Inhalation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Per sponsor request. Closure was not prompted by any safety or efficacy concerns.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3721-II -01
Record Dates: First submitted 2022-03-15; First posted 2022-03-23 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC3721 suspension for inhalation (Experimental): TQC3721 suspension for inhalation, four weeks as a treatment cycle.
  Interventions: Drug: TQC3721 suspension for inhalation
- TQC3721 suspension placebo for inhalation (Placebo Comparator): TQC3721 suspension placebo for inhalation, four weeks as a treatment cycle.
  Interventions: Drug: TQC3721 suspension placebo for inhalation

INTERVENTIONS:
Drug: TQC3721 suspension for inhalation — TQC3721 suspension for inhalation is Dual PDE3/4 inhibitor
  Arms: TQC3721 suspension for inhalation
Drug: TQC3721 suspension placebo for inhalation — TQC3721 suspension for inhalation is Dual PDE3/4 inhibitor
  Arms: TQC3721 suspension placebo for inhalation

SUMMARY:
TQC3721 suspension for inhalation is a PDE3/4 inhibitor developed by Chia Tai Tianqing Pharmaceutical Group Co., LTD., which can simultaneously achieve bronchial smooth muscle relaxation and anti-inflammatory effects. This is a randomized, double-blind, placebo-parallel, phase II trial of the efficacy and safety of inhaled TQC3721 suspension/placebo at different doses in patients with moderate to severe chronic obstructive pulmonary disease. Objective To evaluate the efficacy, safety and tolerability of TQC3721 inhalation suspension in the treatment of moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* 1 Sign the informed consent form before the trial, fully understand the content, process and possible adverse reactions of the test;
* 2 Capable of using the study nebulizer correctly and complying with all study restrictions and procedures;
* 3 Aged between 18 and 75 years old, both men and women;
* 4 Body mass index(BMI)=weight (kg)/height 2 (m2), BMI is 18-28 kg/m2 (including the critical value) and body weight is ≥45kg;
* 5 Subjects have no pregnancy plan and have voluntarily taken effective contraceptive measures for at least 1 month after being screened to the last use of the study drug;
* 6 12-lead electrocardiogram with QT interval corrected ≤450 msec (males) or ≤470 msec (females), QRS interval ≤120 msec, PR interval ≤200 msec and no morphologic and other clinical significant abnormalities that the investigator considered inappropriate for the study;
* 7 Ability to perform acceptable and reproducible spirometry;
* 8 Patients previously treated with LAMA or LABA who had evidence of stable use for at least 3 months prior to screening and agreed to continue use during the study period;
* 9 Capable of withholding LAMA or LABA（ Twice-Daily maintenance LAMA or LABA for at least 24 hours and Once-Daily maintenance LAMA or LABA for at least 48 hours) and SAMA、SABAs（at least 4 hours）prior to initiation of any spirometry;
* 10 According to the 2020 GOLD Guidelines, Post-bronchodilator spirometry at screening must demonstrate FEV1/FVC ratio of ≤0.70 and FEV1 must be ≥30 % to ≤80% of predicted normal;
* 11 Current or former cigarette smokers with a history of cigarette smoking ≥10 pack years (eg, 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years, former cigarette smokers should stop smoke at least 6 months before visit 1).

Exclusion Criteria:

* 1 Intolerance to salbutamol or this product.
* 2 ≥1 hospitalization for COPD treatment within 6 months prior to screening.
* 3 Antibiotic treatment for lower respiratory tract infection within 3 months prior to screening.
* 4 Use of prohibited medications within the time intervals.
* 5 Patients who were currently diagnosed with asthma, active tuberculosis, lung cancer and other active lung diseases and were considered unsuitable for the study.
* 6 Previous lung resection or lung reduction surgery.
* 7 Pulmonary rehabilitation, unless such treatment has been stable from 4 weeks prior to Screening and remains stable during the study.
* 8 A history of drug or alcohol abuse in the past 3 years (14 units of alcohol consumed per week: 1 unit =360 ml of beer or 45 ml of 40% alcohol spirits or 150 ml of wine).
* 9 Have participated in a clinical trial within one month prior to screening or within 5 half-lives of the investigational drug, whichever is the longer.
* 10 Women who are breast-feeding.
* 11 A history of myocardial infarction, congestive heart failure, and unstable or uncontrolled hypertension (systolic blood pressure ≥160mmHg and diastolic blood pressure ≥100mmHg after drug control) within 6 months prior to screening.
* 12 History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localised basal cell carcinoma of the skin.
* 13 Alanine aminotransferase (ALT) or aspartate aminotransferase(AST)≥ 2 x upper limit of normal (ULN), or other abnormal test results were deemed unsuitable for inclusion by the investigator.
* 14 Required use of oxygen therapy, even on an occasional basis.
* 15 Other conditions that the investigator considered inappropriate for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
The peak of Forced Expiratory Volume(FEV1) | From the enrollment of the subjects to four weeks after administration
  Change of the maximum value of FEV1 was determined from baseline to 30minute, 1hour, 2hour and 3hour after medication at week four

SECONDARY OUTCOMES:
Morning trough FEV1 | From the enrollment of the subjects to four weeks after administration
  The FEV1 was determined before administration
Average FEV1 | From the enrollment of the subjects to four weeks after administration
  Average FEV1 twelve hours after administration
COPD Assessment Test (CAT) | From enrollment to four weeks after administration
  Mean Change From Baseline in COPD Assessment Test (CAT) Scoring at Week four. The score range is zero to Fourty points (zero to ten is minor influence; eleven to twenty are moderate; twenty one to thirty are classified as severe impact; thirty one to forty is very severe), and more than ten is more symptoms.
Rescue medication | From baseline to four weeks after administration
  Frequency of Rescue medication use during the study
Incidence of adverse events | from baseline to four weeks after administration
  The Incidence of adverse events as assessed by CTCAE (Common Terminology Criteria for Adverse Events) v5.0
Number of adverse events related to the study drug | from baseline to four weeks after administration
  The number of adverse events associated with the study drug assessed by CTCAE V5.0
Incidence of adverse events associated with the study drug | from baseline to four weeks after administration
  Incidence of adverse events associated with the study drug as assessed by CTCAE V5.0

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - The Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jianxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan